CLINICAL TRIAL: NCT05745103
Title: Optimizing Behavioral Healthcare Delivery Through Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eleos Health (Industry)
Collaborators: Missouri Department of Mental Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: O1Z2A3R4K5
Record Dates: First submitted 2023-02-07; First posted 2023-02-27 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Mood Disorders; Anxiety Disorders
Keywords: Mood Disorders; Anxiety Disorders; Evidence-Based Practices; Community-Based Clinics; Artificial Intelligence
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Open Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Eleos Health Platform (Experimental): Therapists in the AI group will use the HIPAA-compliant, secure, password-protected Eleos Health platform. This AI tool was designed for behavioral health to support clinical decision-making and automation of administrative tasks. The platform captures the therapist and patient's utterances during a treatment session, analyzes the data, and offers feedback on the implementation of EBPs. The platform also incorporates a measurement-based care component, wherein standardized assessment scales completed by clients are immediately summarized and graphed for the therapist, who can use these data to inform therapy and share them with the patient. Insights and key indicators from the session data and MBC are summarized into a progress note draft which the therapist can then submit or edit as needed.
  Interventions: Behavioral: Cognitive behavioral therapy with AI
- Treatment as Usual (Active Comparator): Participants randomized to the control group will receive the routine services provided in the center. Therapists providing TAU will be permitted to use the strategies they deen would be most successful.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy with AI — Cognitive behavioral therapy is a psycho-social intervention that aims to reduce symptoms of various mental health conditions, primarily depression and anxiety disorders. The Eleos Health platform provides real-time data that optimizes this therapy and helps the provider tailor the intervention to the specific client.
  Arms: The Eleos Health Platform
Behavioral: Cognitive behavioral therapy — Cognitive behavioral therapy is a psycho-social intervention that aims to reduce symptoms of various mental health conditions, primarily depression and anxiety disorders.
  Arms: Treatment as Usual

SUMMARY:
The goal of this randomized controlled clinical trial is to determine the feasibility, acceptability, and preliminary efficacy of an artificial intelligence platform )שׁ( for behavioral health in facilitating better clinical outcomes for adult patients receiving outpatient therapy.

The main question[s] it aims to answer are:

* whether an AI platform designed for behavioral healthcare would be feasible and acceptable to patients and therapists.
* whether the depression and anxiety outcomes of adults receiving outpatient cognitive-behavioral therapy (CBT) in a community-based clinic would be superior among patients whose therapists used an AI-based platform to support clinical decision making and administrative tasks compared to patients receiving treatment-as-usual (TAU).

Participants will receive CBT for depression or anxiety and complete standardized assessments. Participants will be followed for the first two months of therapy.

DETAILED DESCRIPTION:
The need for scalable delivery of mental health care services that are efficient and effective is now a major public health priority. Artificial intelligence (AI) tools have the potential to improve behavioral healthcare services by helping clinicians collect objective data on patients' progress, streamline their workflow, and automate administrative tasks.

The goal of this study is to determine the feasibility, acceptability, and preliminary efficacy of an AI platform for behavioral health in facilitating better clinical outcomes for patients receiving outpatient therapy.

This open randomized clinical trial will compare an AI platform provided by Eleos Health to treatment-as-usual (TAU) during the first 2 months of therapy. The study will be conducted at a community-based clinic in the U.S. Participants will be adults referred for outpatient, individual cognitive behavioral therapy for a main diagnosis of a depressive or anxiety disorder. Patients will be randomized to receive either therapy provided with the support of an AI platform developed by Eleos Health or TAU at the same clinic.

Data analysis will be carried out based on intention-to-treat principle. The primary outcomes include the feasibility and acceptability of the AI platform. Secondary outcomes include changes in depression (Patient Health Questionnaire-9) and anxiety (Generalized Anxiety Disorder-7) scores as well as treatment attendance and satisfaction.

Findings of this study will inform the optimization of future trials and services offered to individuals seeking mental health support in the U.S.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old.
2. Presenting for an outpatient CBT for a depressive or anxiety disorder.

Exclusion Criteria:

1. Age <18.
2. individuals who are medically unstable for outpatient treatment.
3. a severe mental health condition that might interfere with treatment compliance (e.g., psychotic depression, psychosis, active substance dependence).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  The PHQ-9 is intended as a tool to assist clinicians with identifying and diagnosing depression.
Patient Health Questionnaire-9 (PHQ-9) | 1 month
  The PHQ-9 is intended as a tool to assist clinicians with identifying and diagnosing depression.
Patient Health Questionnaire-9 (PHQ-9) | 2 months
  The PHQ-9 is intended as a tool to assist clinicians with identifying and diagnosing depression.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline
  The GAD-7 is intended as a tool to assist clinicians with identifying and diagnosing anxiety.
Generalized Anxiety Disorder-7 (GAD-7) | 1 month
  The GAD-7 is intended as a tool to assist clinicians with identifying and diagnosing anxiety.
Generalized Anxiety Disorder-7 (GAD-7) | 2 months
  The GAD-7 is intended as a tool to assist clinicians with identifying and diagnosing anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ozark Center, Joplin, Missouri, United States

REFERENCES:
- [Background] Peretz G, Taylor CB, Ruzek JI, Jefroykin S, Sadeh-Sharvit S. Machine Learning Model to Predict Assignment of Therapy Homework in Behavioral Treatments: Algorithm Development and Validation. JMIR Form Res. 2023 May 15;7:e45156. doi: 10.2196/45156. PMID 37184927
- [Background] Kellogg KC, Sadeh-Sharvit S. Pragmatic AI-augmentation in mental healthcare: Key technologies, potential benefits, and real-world challenges and solutions for frontline clinicians. Front Psychiatry. 2022 Sep 6;13:990370. doi: 10.3389/fpsyt.2022.990370. eCollection 2022. PMID 36147984
- [Background] Sadeh-Sharvit S, Rego SA, Jefroykin S, Peretz G, Kupershmidt T. A Comparison Between Clinical Guidelines and Real-World Treatment Data in Examining the Use of Session Summaries: Retrospective Study. JMIR Form Res. 2022 Aug 16;6(8):e39846. doi: 10.2196/39846. PMID 35972782
- [Result] Sadeh-Sharvit S, Camp TD, Horton SE, Hefner JD, Berry JM, Grossman E, Hollon SD. Effects of an Artificial Intelligence Platform for Behavioral Interventions on Depression and Anxiety Symptoms: Randomized Clinical Trial. J Med Internet Res. 2023 Jul 10;25:e46781. doi: 10.2196/46781. PMID 37428547